CLINICAL TRIAL: NCT01913717
Title: Short-term High Precision Radiotherapy for Early Prostate Cancer With Concomitant Boost on the Dominant Lesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO S768/113; 2012-IG133218 (Other Grant/Funding Number: AIRC)
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Adenocarcinoma of Prostate
Keywords: Prostate cancer; Radiotherapy; hypofractionated radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- External beam radiotherapy (Experimental): External beam radiotherapy
  Interventions: Radiation: External beam radiotherapy

INTERVENTIONS:
Radiation: External beam radiotherapy — The patients will be treated with extreme hypofractionated radiotherapy with the dose delivery system that will result most fit at the in-silica study. Simultaneous Integrated Boost (SIB) technique will be applied to deliver a total dose of 36.25 Gy in 5 fractions (over 10 days) to the whole prostate (7.25 Gy/fraction) and 37.5 Gy to the dominant intraprostatic lesion DIL (7.5 Gy/fraction), profiting of the high sensibility of prostate cancer to high dose/fraction. Several strategies will be applied in order to reduce the dose to the surrounding organs at risk.
  Other Names: hypofractionated radiotherapy

SUMMARY:
The present research project aims to improve the current treatment for prostate-confined tumor, evaluating the safety and feasibility of a very short hypofractionated radiotherapy schedule administered with one of the best available dose delivery systems. The study will include 2 sub-studies (in-silica and clinical study) and 4 tasks.

DETAILED DESCRIPTION:
Approximately 70% of men with newly diagnosed prostate cancer feature organ-confined disease. Conventional treatment options for prostate-confined cancer include radical prostatectomy, external beam radiation therapy, brachytherapy and active surveillance. All currently available treatments have comparable toxicity risk and high social and economic impact, hence the best treatment option has not been defined yet. In the radiation oncology field the gold standard for prostate cancer management is 7-8 weeks intensity modulated radiotherapy (IMRT), which can be delivered with the latest generation of accelerators providing modulated arc delivery (eg. RapidArc™, Varian) or with newly developed machines such as the Vero system (BrainLab AG - Mitsubishi Heavy Industries Ltd). The present research project aims to improve the current treatment for prostate confined tumor, evaluating the best strategy to deliver a very-short hypofractionated radiotherapy scheme. In the first part of this AIRC grant an in-silica study will be performed on 10 test prostate cancer patients, with comparative competitive treatment plans with the state of the art treatment options for prostate cancer: the Vero system, the RapidArc system, the Cyberknife (all available at the European Institute of Oncology IEO, Milan, Italy), and protontherapy (available at the Centre of Adrotherapy, in Pavia, Italy). This dosimetric comparison will be performed in order to define the technique that provides the maximum target coverage with the minimum dose to the surrounding organs at risk (OARs) to be used to perform the clinical trial that will follow within this AIRC grant. After performing the in-silica study, 65 newly diagnosed prostate cancer patients with 2011 National Comprehensive Cancer Network (NCCN) risk category ranging from very low to intermediate but not undergoing hormonal treatment, will be consecutively enrolled in a prospective phase II trial. The patients will be treated at the Division of Radiation Oncology of the IEO, with the dose delivery system that will result most fit at the in-silica study. Simultaneous Integrated Boost (SIB) technique will be applied to deliver a total dose of 36.25 Gy in 5 fractions (over 10 days) to the whole prostate (7.25 Gy/fraction) and 37.5 Gy to the dominant intraprostatic lesion DIL (7.5 Gy/fraction), profiting of the high sensibility of prostate cancer to high dose/fraction. Several strategies will be applied in order to reduce the dose to the surrounding OARs. In order to define the localization of the DIL, multiparametic magnetic resonance imaging (MRI) of the pelvis will be performed (with spectroscopy, diffusion weighted and perfusion acquisitions), and fused with computed tomography (CT) scan. In-room image-guidance will be applied at each treatment section, in order to minimize uncertainties in intra and inter-fraction prostate localization. At the end of the radiotherapy course, each patient will be followed-up, in order to assess the treatment safety and effectiveness in terms of early and late toxicity, and tumor control. A sampling from the prostate tumor tissue for biological study will be taken for microarray analysis. The expression of specific markers of radiosensitivity and radioresistance will be investigated.

ELIGIBILITY:
Inclusion Criteria:

- Histologically confirmed adenocarcinoma of prostate, including the following 2011 National Comprehensive Cancer Network (NCCN) risk categories: very low (T1c PSA <10 ng/ml, Gleason score <7, fewer than 3 positive biopsy cores, <50% cancer in each core, PSA density <0.15 ng/ml) or low (T1-T2a, PSA <10 ng/ml, Gleason score <7) or intermediate (T2b or T2c, PSA between 10 and 20 ng/ml, Gleason score of 7)

* cN0 and cM0 stage
* Age > 18 years
* Good performance status (ECOG< 2),
* No previous pelvic radiotherapy
* No previous prostatectomy
* No hormonal treatment (neoadjuvant or concomitant)
* No concomitant bowel inflammatory disease or other serious comorbidities
* Good urinary flow (peak flow > 10 ml/s)
* No previous invasive cancer (within 5 years before the prostate cancer diagnosis) apart from non-melanoma skin malignancies.

Exclusion Criteria:

* Extraprostatic tumor extension (T3) or locally advanced disease (T4)
* Pelvic lymph node metastasis (N1)
* Distant metastasis (M1)
* Urinary obstructive symptoms (IPSS > 20)
* Previous pelvic radiotherapy
* Severe systemic disorders
* Concomitant disorders including: chronic urinary or intestinal inflammatory conditions (for example, ulcerous recto-colitis, Crohn disease), anti-coagulant treatment (warfarin, heparin)
* Previous malignancy except for skin non-melanoma cancer or 3-year disease free interval from previous malignancy like in situ cervix cancer or non muscle invasive bladder cancer
* Non conformity of the radiotherapy dose distribution when compared to the dose constraints
* Psychiatric disorders or any other condition that can can make unreliable the informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | one month after radiotherapy
  The primary outcome is the acute toxicity according to the validated scale Radiotherapy Oncology Group / European Organization for Research and Treatment of Cancer (RTOG / EORTC). It will measure the proportion of patients who experience at least one event of acute toxicity of grade 3 or 4 according to the scale RTOG / EORTC) as the maximum value of toxicity during radiation treatment or within one month after the completion of radiotherapy.

SECONDARY OUTCOMES:
late toxicity | 2 years
  late toxicity according to Scala CTCAE v4.0 toxicity criteria and scale RTOG / EORTC
efficacy of treatment | 2 years
  assessed in terms of
  * biochemical progression free survival (biochemical relapse, i.e. rising PSA)
  * pattern of relapse
  * clinical progression free survival (including local or distant recurrence)
  * overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Orecchia, MD, Principal Investigator — European Institute of Oncology; BARBARA A JERECZEK, MD PhD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Corrao G, Marvaso G, Zaffaroni M, Volpe S, Augugliaro M, Fodor CI, Zerini D, Vingiani A, Mistretta FA, Luzzago S, Alessi S, Pricolo P, Musi G, De Cobelli O, Renne G, Manzoni M, Petralia G, Orecchia R, Jereczek-Fossa BA. Correlation between radiological and biological features and clinical outcomes in early prostate cancer: an exploratory subgroup analysis. Neoplasma. 2022 Mar;69(2):404-411. doi: 10.4149/neo_2021_210622N828. Epub 2022 Jan 12. PMID 35014537
- [Derived] Marvaso G, Ciardo D, Gandini S, Riva G, Frigo E, Volpe S, Fodor C, Zerini D, Rojas DP, Comi S, Cambria R, Cattani F, Musi G, De Cobelli O, Orecchia R, Jereczek-Fossa BA. Comparison of Outcomes and Toxicity Between Extreme and Moderate Radiation Therapy Hypofractionation in Localized Prostate Cancer: A Propensity Score Analysis. Int J Radiat Oncol Biol Phys. 2019 Nov 15;105(4):735-744. doi: 10.1016/j.ijrobp.2019.07.027. Epub 2019 Aug 1. PMID 31377161
- [Derived] Cremonesi M, Garibaldi C, Timmerman R, Ferrari M, Ronchi S, Grana CM, Travaini L, Gilardi L, Starzynska A, Ciardo D, Orecchia R, Jereczek-Fossa BA, Leonardi MC. Interim 18F-FDG-PET/CT during chemo-radiotherapy in the management of oesophageal cancer patients. A systematic review. Radiother Oncol. 2017 Nov;125(2):200-212. doi: 10.1016/j.radonc.2017.09.022. Epub 2017 Oct 10. PMID 29029833
- [Derived] Garibaldi C, Ronchi S, Cremonesi M, Gilardi L, Travaini L, Ferrari M, Alterio D, Kaanders JHAM, Ciardo D, Orecchia R, Jereczek-Fossa BA, Grana CM. Interim 18F-FDG PET/CT During Chemoradiation Therapy in the Management of Head and Neck Cancer Patients: A Systematic Review. Int J Radiat Oncol Biol Phys. 2017 Jul 1;98(3):555-573. doi: 10.1016/j.ijrobp.2017.02.217. Epub 2017 Mar 4. PMID 28581396
- [Derived] Jereczek-Fossa BA, Fanetti G, Fodor C, Ciardo D, Santoro L, Francia CM, Muto M, Surgo A, Zerini D, Marvaso G, Timon G, Romanelli P, Rondi E, Comi S, Cattani F, Golino F, Mazza S, Matei DV, Ferro M, Musi G, Nole F, de Cobelli O, Ost P, Orecchia R. Salvage Stereotactic Body Radiotherapy for Isolated Lymph Node Recurrent Prostate Cancer: Single Institution Series of 94 Consecutive Patients and 124 Lymph Nodes. Clin Genitourin Cancer. 2017 Aug;15(4):e623-e632. doi: 10.1016/j.clgc.2017.01.004. Epub 2017 Jan 11. PMID 28185875
- [Derived] Timon G, Ciardo D, Bazani A, Garioni M, Maestri D, De Lorenzo D, Pansini F, Cambria R, Rondi E, Cattani F, Marvaso G, Zerini D, Vischioni B, Ciocca M, Russo S, Molinelli S, Golino F, Scroffi V, Rojas DP, Fodor C, Petralia G, Santoro L, De Cobelli O, Orecchia R, Jereczek-Fossa BA. Rationale and protocol of AIRC IG-13218, short-term radiotherapy for early prostate cancer with concomitant boost to the dominant lesion. Tumori. 2016 Oct 13;102(5):536-540. doi: 10.5301/tj.5000547. Epub 2016 Aug 5. PMID 27514314
- See also: AIRC: ASSOCIAZIONE ITALIANA PER LA RICERCA SUL CANCRO — http://www.airc.it